CLINICAL TRIAL: NCT01650818
Title: Exercise traiNing in Amyotrophic Lateral Sclerosis: a ranDomized Trial Comparing Home-based Aerobic endUrance tRAiNing vs. Usual physiCal Therapy intErvention
Brief Title: Aerobic Exercise Training in Amyotrophic Lateral Sclerosis
Acronym: ENDURANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Alessandro Mezzani, MD, FESC, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEC641
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Aerobic training; Peak oxygen consumption; Quality of life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise training (Experimental)
  Interventions: Other: Aerobic exercise training
- Standard physical therapy (Active Comparator)
  Interventions: Other: Standard physical therapy (Stretching/Range-of-motion)

INTERVENTIONS:
Other: Aerobic exercise training — Intensity: heart rate corresponding to 40% peak VO2. Frequency: 5 sessions/week. Duration: 5 min warm-up + 20 min training + 5 min cool-down during the 1st month; 5 min warm-up + 30 min training + 5 min cool-down during the 2nd and 3rd month
  Arms: Aerobic exercise training
Other: Standard physical therapy (Stretching/Range-of-motion) — Intensity: N/A. Frequency: 5 sessions/week. Duration: 5 min warm-up + 20 min training + 5 min cool-down during the 1st month; 5 min warm-up + 30 min training + 5 min cool-down during the 2nd and 3rd month
  Arms: Standard physical therapy

SUMMARY:
The purpose of this study is to compare the safety and the effects of moderate-intensity aerobic endurance training to those of an usual physical therapy intervention on exercise capacity and quality of life in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Scarce evidence is available regarding aerobic exercise training of patients with ALS. Some studies using transgenic mouse models of familial ALS have shown markedly slowed disease progression, improved functional capacity, and extension of survival in animals undergoing aerobic exercise training. In humans, only one non-randomized study has shown that moderate-intensity aerobic exercise training was of little beneficial effect in a small group of patients with Kennedy disease, a rare X-linked progressive neuromuscular disease involving lower motorneurons, presenting a pathophysiological picture quite different from that of ALS. To the best of our knowledge, the safety and the effects of aerobic exercise training on functional capacity and quality of life of patients with ALS have not been systematically evaluated as yet in a randomized, controlled trial with an adequate sample size.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite ALS, probable ALS, or probable-laboratory supported ALS according to the El Escorial criteria or diagnosis of progressive muscular atrophy.
* Ability to perform a baseline symptom-limited cardiopulmonary exercise test with attainment of peak power and respiratory exchange ratio of >= 50 W and >= 1.00, respectively.
* Time since symptoms onset <= 18 months.
* Forced vital capacity >= 70% of predicted.
* Informed written consent.

Exclusion Criteria:

* Coexisting neurological disease.
* Coexisting extra-neurological disease significantly affecting exercise capacity.
* Coexisting malignancy.
* Ongoing/planned pregnancy.
* Involvement in formal endurance and/or strength training program.
* Enrolment in any other clinical trial.
* Cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in peak oxygen consumption (peak VO2) | 3 months
  Evaluate the effects of aerobic training on peak VO2, as assessed by cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Aerobic training safety and tolerability | 3 months
  Evaluate aerobic training safety and tolerability in terms of adverse events incidence and adherence to training program
Change from baseline in quality of life | 3 months
  Evaluate the effects of aerobic training on quality of life, as assessed by McGill questionary
Change from baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) score | 3 months
  Evaluate the effects of aerobic training on the ALSFRS-R score
Change from baseline in lower limbs muscle strength | 3 months
  Evaluate the effects of aerobic training on isometric muscle strength of lower limbs, as assessed by isometric dynamometry
Change from baseline in upper and lower motor neurons function at the upper and lower limbs level | 3 months
  Evaluate the effects of aerobic training on upper and lower motor neurons function at the upper and lower limbs level, as determined by compound muscle action potential and neurophysiological index and motor evoked potentials
Change from baseline in ventilatory function | 3 months
  Evaluate the effects of aerobic training on ventilatory function, as assessed by spirometry and measurement of maximal inspiratory and expiratory pressures
Change from baseline in circulating inflammatory markers, growth factors and descriptors of skeletal muscle damage | 3 months
  Evaluate the effects of aerobic training on circulating inflammatory markers and growth factors (CRP, TNF-alfa, IL-6, Angiogenin, Angiopoietin 1 and 2, Thrombospondin, VEGF, BDNF, IGF-1) and markers of skeletal muscle damage (CPK)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Mezzani, MD, Principal Investigator — Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Veruno; Fabrizio Pisano, MD, Study Director — Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Veruno
Locations (1):
- Fondazione Salvatore Maugeri, IRCCS - Scientific Institute of Veruno, Veruno, Italy

REFERENCES:
- [Background] Mezzani A, Pisano F, Cavalli A, Tommasi MA, Corra U, Colombo S, Grassi B, Marzorati M, Porcelli S, Morandi L, Giannuzzi P. Reduced exercise capacity in early-stage amyotrophic lateral sclerosis: Role of skeletal muscle. Amyotroph Lateral Scler. 2012 Jan;13(1):87-94. doi: 10.3109/17482968.2011.601463. Epub 2011 Aug 11. PMID 21830991